CLINICAL TRIAL: NCT00270530
Title: Intermittent Preventive Treatment of Malaria With Sulfadoxine-Pyrimethamine in HIV-Seropositive and HIV-Seronegative Pregnant Women in Zambia
Brief Title: Intermittent Preventive Treatment of Malaria in HIV-Seropositive Pregnant Women in Zambia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center for International Health and Development (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: S1954-21/22-2
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2006-01-31 (Estimated); Status verified 2004-11

CONDITIONS: Placental Malaria Infection; HIV Infections; Stillbirth; Prematurity; Neonatal Deaths
Keywords: Malaria; Placental diseases; Birth complications; Plasmodium falciparum; Zambia; HIV-seropositive; HIV
MeSH Terms: conditions — HIV Infections; Stillbirth; Premature Birth; Perinatal Death; Malaria; Placenta Diseases; Malaria, Falciparum; HIV Seropositivity | interventions — fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine (Fansidar)

SUMMARY:
Prevention of malaria in pregnancy is critical given the high incidence of malaria in Zambia and its serious impact on both maternal and infant survival. Intermittent presumptive treatment with sulfadoxine-pyrimethamine has been shown to be highly efficacious for reducing the risk of malaria in pregnancy. However, based on a study done in western Kenya, HIV-infected pregnant women may need more frequent dosing of SP, i.e., on a monthly basis rather than the standard 2-dose regimen given during the second and third trimesters, as HIV appears to reduce the effectiveness of the SP drug combination. The goal of this study was to evaluate the efficacy of the standard dosing regimen in comparison to an intensive monthly SP dosing schedule in HIV-positive women.

DETAILED DESCRIPTION:
Primary Objectives

To compare the efficacy of IPT with monthly SP versus a two-dose regimen given once in the second and once in the third trimester in HIV-infected women on the:

* Prevalence of placental malaria infection
* Prevalence of maternal peripheral parasitemia

Secondary objectives

To compare IPT with monthly SP versus a two-dose regimen given once in the second and once in the third trimester in HIV-infected women on:

* Birth weight, including the proportion of LBW infants
* Incidence of prematurity
* Neonatal and fetal death and third trimester stillbirth
* Incidence of neonatal jaundice
* Third trimester anemia
* Third trimester severe anemia
* Proportion of mothers who develop symptomatic malaria during the course of pregnancy

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive pregnant women between 16-28 weeks of gestation identified through VCT
* HIV-negative pregnant women between 16-28 weeks of gestation identified through VCT
* Residence within the catchment area of the health facility
* Willing to deliver at the health facility
* Willing to agree to adhere to the requirements of study participation (including monthly ANC visits and willing to allow all study procedures)
* Willing to provide written informed consent
* Aged 18 years and above

Exclusion Criteria:

* Severe anemia (Hb < 6 g/dL)
* History of allergic reactions to sulfa drugs
* History of known pregnancy complications (e.g. breech presentation, severe pre-eclampsia, prior caesarian section)
* History or presence of major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis, prior to randomization
* Any significant presenting illness that requires hospitalization
* Intent to move out of the study catchment area before delivery or deliver at relative's home out of the catchment area
* Prior enrollment in the study or concurrent enrollment in another study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 454
Dates: Start 2002-11; Study Completion 2004-10

PRIMARY OUTCOMES:
• Prevalence of placental malaria infection
• Prevalence of maternal peripheral parasitemia

SECONDARY OUTCOMES:
• Prevalence of maternal peripheral parasitemia
• Birth weight, including the proportion of LBW infants
• Incidence of prematurity
• Neonatal and fetal death and third trimester stillbirth
• Incidence of neonatal jaundice
• Third trimester anemia
• Third trimester severe anemia
• Proportion of mothers who develop symptomatic malaria during the course of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Davidson H Hamer, MD, Principal Investigator — Center for International Health and Development, Boston University
Locations (1):
- Tropical Diseases Research Centre, Ndola, Zambia

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Hamer DH, Mwanakasale V, Macleod WB, Chalwe V, Mukwamataba D, Champo D, Mwananyanda L, Chilengi R, Mubikayi L, Mulele CK, Mulenga M, Thea DM, Gill CJ. Two-dose versus monthly intermittent preventive treatment of malaria with sulfadoxine-pyrimethamine in HIV-seropositive pregnant Zambian women. J Infect Dis. 2007 Dec 1;196(11):1585-94. doi: 10.1086/522142. Epub 2007 Oct 25. PMID 18008241